CLINICAL TRIAL: NCT01934075
Title: Development of Mental Health Treatment for Obstetric Fistula Patients in Tanzania
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH); Kilimanjaro Christian Medical Centre, Tanzania (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: R21HD073681 (NIH); R21HD073681 (NIH)
Record Dates: First submitted 2013-08-29; First posted 2013-09-04 (Estimated); Last update posted 2016-08-09 (Estimated); Status verified 2016-08

CONDITIONS: Other Obstetric Trauma OS
Keywords: Obstetric fistula; Mental health; Tanzania
MeSH Terms: conditions — Psychological Well-Being

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Mental health treatment (Experimental): Participants will receive twice-weekly exposure to 6 sessions of individual mental health treatment in a private room. Sessions will follow the intervention manual and be delivered by a full-time nurse facilitator who has a counseling background and receives supervision by a trained therapist.
  Interventions: Behavioral: Mental health treatment
- Standard of Care (No Intervention): Participants in the control condition will receive counseling that is the current standard of care for fistula patients at KCMC.

INTERVENTIONS:
Behavioral: Mental health treatment — 6 sessions of individual mental health counseling.
  Arms: Mental health treatment

SUMMARY:
The purpose of this study is to determine whether a mental health intervention for obstetric fistula patients in Tanzania improves primary outcomes (depression, PTSD and somatic symptoms) and secondary outcomes (coping, perceived stigma, social support, social participation, efficacy to engage with providers, adherence to clinical recommendations and social reintegration).

DETAILED DESCRIPTION:
Obstetric fistula is a hole between the bladder or rectum and the vagina, which develops when obstructed labor is not relieved by cesarean section and results in uncontrollable leaking of urine and/or feces. The only cure for obstetric fistula is surgical repair. Multiple studies have documented the social and psychological impact of obstetric fistula, which includes social isolation, stigma, depression, and mental health dysfunction. The surgical repair setting can be a window of opportunity to address the accumulated mental health distress of living with a fistula. However, to date no intervention studies have evaluated empirically-supported therapies to assist in psychological healing among fistula patients. The proposed study aims to fill this gap by developing and pilot-testing a theoretically informed mental health intervention for women receiving surgical repair for obstetric fistula at KCMC Hospital in Moshi, Tanzania. The study has three specific aims: 1) To develop the nurse-delivered mental health intervention, built on theories of coping and cognitive behavioral therapy, 2) To assess feasibility and acceptability of implementing the intervention in the KCMC fistula ward, considering: intervention fidelity, patient satisfaction, provider feedback and cost of delivery, 3) To assess effectiveness of the intervention by comparing immediate and short term outcomes in 30 women who receive the experimental intervention with 30 women receiving the standard of care counseling, examining differences in primary outcomes (depression, PTSD and somatic symptoms) and secondary outcomes (coping, perceived stigma, social support, social participation, efficacy to engage with providers, adherence to clinical recommendations and social reintegration). The proposed research directly responds to the needs specified by NIH because it expands the "evidence base for improving social outcomes" of women with obstetric fistula and develops a "sustainable intervention" that complements existing local care (PA-11-143). At the completion of this study, it is our expectation that we will have a structured intervention curriculum and supportive preliminary data to inform an R01 application to conduct a multi-site evaluation of the intervention, which, if effective, can be disseminated to fistula repair clinics internationally.

ELIGIBILITY:
Inclusion Criteria:

* Patients at the Kilimanjaro Christian Medical Center Obstetrics-Gynecology Department, receiving surgical repair for a fistula resulting from childbirth

Exclusion Criteria:

* Impaired mental status

Ages: 18 Years to 99 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2013-09; Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Depression symptoms | 90 days
  Self-report, measured by Center for Epidemiological Studies Depression Scale (CES-D)

SECONDARY OUTCOMES:
PTSD symptoms | 90 days
  Self-report, measured by the PTSD Checklist, civilian version
Anxiety symptoms | 90 days
  Self-report, measured by the Beck Anxiety Inventory

CONTACTS AND LOCATIONS:
Overall Officials: Melissa Watt, PhD, Principal Investigator — Duke University
Locations (1):
- Kilimanjaro Christian Medical Center, Moshi, Tanzania

IPD SHARING:
Plan to Share IPD: Yes
Data will be made available upon request.

REFERENCES:
- [Derived] Watt MH, Mosha MV, Platt AC, Sikkema KJ, Wilson SM, Turner EL, Masenga GG. A nurse-delivered mental health intervention for obstetric fistula patients in Tanzania: results of a pilot randomized controlled trial. Pilot Feasibility Stud. 2017 Sep 12;3:35. doi: 10.1186/s40814-017-0178-z. eCollection 2017. PMID 28912958